CLINICAL TRIAL: NCT06303830
Title: Changes Induced by Bariatric Surgery in Cardiovascular Responses to Dietary Supplementation With Sodium Nitrate
Brief Title: Bariatric Surgery and Cardiovascular Responses to Sodium Nitrate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Jéssica Maria Sanches Lopes, PhD in Pharmacology, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BACA2019
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — sodium nitrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Sodium nitrate, once a day for 14 days
  Interventions: Dietary Supplement: Sodium nitrate
- Bariatric group (Experimental): Sodium nitrate, once a day for 14 days
  Interventions: Dietary Supplement: Sodium nitrate

INTERVENTIONS:
Dietary Supplement: Sodium nitrate — Sodium Nitrate

SUMMARY:
Inorganic nitrite and nitrate can be reduced to NO and NO-related species such as S-nitrosothiols via the nitrate-nitrite-NO pathway. This is due to the reduction of nitrate to nitrite by the action of bacteria in the mouth and the reduction of nitrite to NO depending on the acidic pH on the stomach or by enzymes with nitrite-reductase activity. The acidic environment of the stomach is very important to the formation of NO and S-nitrosothiols and several studies suggest that changes in gastric pH can affect this conversion. In this context, bariatric surgery, by altering the anatomy of the stomach and increasing gastric pH, can affect the nitrate-nitrite-NO pathway and change the antihypertensive and antioxidant effect of sodium nitrate.

ELIGIBILITY:
Inclusion Criteria:

* For volunteers who underwent bariatric surgery:

  1. Female;
  2. Age over 18 years old and under 60 years old;
  3. Having had bariatric surgery more than 1 and a half years ago;
  4. Present stabilized weight loss;
* For voluntary controls:

  1. Female;
  2. Age over 18 years old and under 60 years old;

Exclusion Criteria:

* For volunteers who underwent bariatric surgery and controls:

  1. Having uncontrolled blood pressure (above 160/100 mmHg), even with use regulate up to two antihypertensive agents;
  2. Hypertensive patients must be using a maximum of two antihypertensives;
  3. Have Diabetes Mellitus or other endocrinopathy;
  4. Have kidney or liver failure;
  5. Individuals who smoke.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Assess changes in s-nitrosothiols | 14 days
  Change in s-nitrosothiols concentration in plasma After Sodium Nitrate Treatment

SECONDARY OUTCOMES:
Assess changes in blood pressure | 14 days
  Change in Blood Pressure After Sodium Nitrate Treatment by Ambulatory blood pressure monitors (ABPMs)
Assess changes in endotelial function | 14 days
  Change in endotelial function After Sodium Nitrate Treatment by Endopat
Assess changes in Vascular stiffness | 14 days
  Change in Vascular stiffness After Sodium Nitrate Treatment by pulse wave velocity (PWV)
Assess changes in nitrate concentration | 14 days
  Change in nitrate concentration in plasma After Sodium Nitrate Treatment
Assess changes in nitrite concentration | 14 days
  Change in nitrite concentration in plasma After Sodium Nitrate Treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Usp - Hospital Das Clínicas Da Faculdade de Medicina de Ribeirão, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No